CLINICAL TRIAL: NCT07167862
Title: Optimizing Preeclampsia Postpartum With Point-of-Care Ultrasound: A Pilot Prospective Cohort Study
Brief Title: Optimizing Preeclampsia Postpartum With Point-of-care Ultrasound
Acronym: PPPOCUS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Ashten B Waks, Assistant Clinical Professor, University of California, Irvine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7178
Record Dates: First submitted 2025-08-15; First posted 2025-09-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Preeclampsia; Preeclampsia Postpartum; Preeclampsia Severe or Mild
Keywords: Preeclampsia; Postpartum; Point of care ultrasound; Diuretics
MeSH Terms: conditions — Pre-Eclampsia; Lymphoma, Follicular | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Cohort 1: POCUS-guided subjects receiving oral furosemide (Experimental): A prospective cohort of patients diagnosed with preeclampsia who will be enrolled and undergo POCUS within 24 hours of delivery. Those meeting pre-specified hemodynamic criteria (> 3 B-lines, maximum IVC diameter > 2 cm, and/or IVC collapsibility index < 15%) will receive a 5-day course of oral furosemide 20mg and oral potassium chloride 40mEq daily.
  Interventions: Diagnostic Test: Butterfly iQ3 ultrasound system for determination of postpartum volume status; Drug: Oral furosemide
- Cohort 2: POCUS-guided subjects receiving intravenous furosemide (Experimental): A prospective cohort of patients diagnosed with preeclampsia who will be enrolled and undergo POCUS within 24 hours of delivery. Those meeting pre-specified hemodynamic criteria (> 3 B-lines, maximum IVC diameter > 2 cm, and/or IVC collapsibility index < 15%) will receive a single dose of intravenous furosemide 40mg and oral potassium chloride 40mEq.
  Interventions: Diagnostic Test: Butterfly iQ3 ultrasound system for determination of postpartum volume status; Drug: Intravenous furosemide
- Cohort 3: Historical matched controls (Active Comparator): A retrospective cohort comprised of patients who delivered before implementation of POCUS-guided postpartum management of preeclampsia (1/1/2024 - 6/1/2025). These patients will be selected from the electronic medical record and matched to enrolled patients for variables such as age, body mass index, gestational age at delivery, severity of preeclampsia, and mode of delivery.
  Interventions: Drug: Oral furosemide; Drug: Intravenous furosemide

INTERVENTIONS:
Diagnostic Test: Butterfly iQ3 ultrasound system for determination of postpartum volume status — A trained study staff member will perform point-of-care ultrasound (POCUS) of the lungs and the inferior vena cava (IVC). All POCUS assessments will be performed using either the curvilinear or phased array settings on a portable Butterfly iQ3 ultrasound system. Images obtained via the Butterfly iQ3 ultrasound system will be labeled according to the subject's unique identification number and transmitted directly to a digital study archive. The lead investigator or physician of record will review all captured ultrasound images to ensure that an appropriate therapy is selected moving forward.
  Any subject who is confirmed to have 3 or more B-lines, a maximum IVC diameter above 2.0cm, or an IVC collapsibility index less than 15% on POCUS will become a candidate for diuretic therapy, which will be ordered by the patient's primary inpatient provider.
  Arms: Cohort 1: POCUS-guided subjects receiving oral furosemide; Cohort 2: POCUS-guided subjects receiving intravenous furosemide
Drug: Oral furosemide — Any subject who is confirmed to have 3 or more B-lines, a maximum IVC diameter above 2.0cm, or an IVC collapsibility index less than 15% on POCUS will become a candidate for diuretic therapy, which will be ordered by the patient's primary inpatient provider. The first cohort of 48 patients will be treated with oral furosemide 20mg daily and oral potassium chloride 40mEq daily for a total of 5-days. As patients delivered vaginally are typically discharged 2-3 days after birth and delivered via cesarean are typically discharged 4-5 days after birth, patients who have not yet completed the medication course by the time of planned discharge will be prescribed the remainder of their medications before departing the hospital.
  Other Names: Oral Lasix
  Arms: Cohort 1: POCUS-guided subjects receiving oral furosemide; Cohort 3: Historical matched controls
Drug: Intravenous furosemide — Any subject who is confirmed to have 3 or more B-lines, a maximum IVC diameter above 2.0cm, or an IVC collapsibility index less than 15% on POCUS will become a candidate for diuretic therapy, which will be ordered by the patient's primary inpatient provider. The second cohort of 48 patients will be treated with a single dose of intravenous furosemide 40mg and oral potassium chloride 40mEq on postpartum day 1.
  Other Names: Intravenous Lasix
  Arms: Cohort 2: POCUS-guided subjects receiving intravenous furosemide; Cohort 3: Historical matched controls

SUMMARY:
This study explores a novel approach to improving care for postpartum patients with preeclampsia, a pregnancy-related condition characterized by high blood pressure, protein in the urine, and organ dysfunction. Preeclampsia affects up to 9% of pregnancies and can progress to include complications of seizures, stroke, and even death. Over 60% of patients with preeclampsia continue to experience high blood pressure at the time of discharge from their delivery hospitalization, and many of these patients require blood pressure medications for up to 6 months postpartum. Even with blood pressure medications, many of these patients are readmitted to the hospital within six weeks of delivery.

In this study, the investigators will utilize point-of-care ultrasound (POCUS), a quick and non-invasive, bedside imaging strategy, to look for signs of excess fluid accumulating in the lungs and venous system of postpartum patients with preeclampsia. Because excess fluid has the potential to worsen blood pressure, subjects with evidence of this on POCUS would be treated with a diuretic medication called furosemide (either orally or intravenously) within 24 hours of delivery.

The investigators' main goal is to determine whether using POCUS can help physicians make better treatment decisions and improve short-term outcomes for postpartum patients with preeclampsia. The investigators' aim to achieve faster recovery of blood pressure, reduce the need for blood pressure medication at hospital discharge, and lower the rates of hospital readmission for those with preeclampsia. This study could significantly enhance the overall care and health of postpartum patients.

DETAILED DESCRIPTION:
Preeclampsia is a condition of the antenatal and postpartum periods, which manifests as new-onset hypertension and proteinuria. Globally, preeclampsia is estimated to affect up to 9% of all pregnancies, though as many as 63% of patients who receive this diagnosis will remain hypertensive beyond the time of postpartum hospital discharge. Because of this, up to 36% of patients with preeclampsia will require antihypertensive therapy at the time of hospital discharge, and between 26 - 74% of patients with preeclampsia will be readmitted during the first six weeks' postpartum. Cumulatively, these preeclampsia-related outcomes result in United States medical expenditures exceeding $36 million annually.

One proposed strategy for improving outcomes among patients with preeclampsia is postpartum administration of diuretics. This treatment is posited to target preeclampsia-related volume overload, which in turn is thought to contribute to continued hypertension in the postpartum period. The earliest trial on the use of diuretics for this purpose was published by Ascarelli et al in 2005 and involved randomization of 264 postpartum patients with preeclampsia to either a 5-day course of oral furosemide 20mg daily or standard preeclampsia management. Outcomes from this study included blood pressure changes over the postpartum hospital stay, need for antihypertensive therapy during hospitalization and at discharge, length of postpartum hospital stay, and other postpartum complications. While this intervention lowered systolic blood pressure by over 10 mm Hg in the first 48 hours postpartum, it did not result in a statistically significant decrease in antihypertensive therapy requirements, postpartum length of stay, or the frequency of other postpartum complications. As recently as 2021, Perdigao and colleagues published the FoR BP trial, which similarly randomized 384 postpartum patients with hypertensive disorders of pregnancy to either a 5-day course of oral furosemide 20mg daily or standard preeclampsia management. Primary outcomes from this study were slightly different from the Ascarelli et al study and included persistent hypertension 7 days postpartum and days to resolution of hypertension. Ultimately, Perdigao et al's results were more promising and demonstrated that a brief course of oral diuretics reduced the incidence of persistent hypertension by nearly 60% in patients with hypertensive disorders of pregnancy.

A potential explanation for this discrepancy in findings from earlier studies is that volume overload affects only a subset of patients with preeclampsia. While preeclamptic patients with volume overload are likely to demonstrate a meaningful response to diuresis, those without significant volume overload are less likely to respond to this treatment. Because the aforementioned studies did not account for patients' volume status at the time of randomization or diuretic administration, it seems possible that they did not sufficiently capture the patient population most likely to respond to the intervention of interest.

With regards to evaluating postpartum volume status and how it might relate to diuretic response, most obstetric practitioners currently rely on findings from physical examination (e.g. jugular venous distension, rales on lung exam, peripheral edema) that are known to have limited sensitivity. However, there is increasing evidence in the obstetric literature that use of POCUS might be a helpful adjunct for determining postpartum volume status. In 2023, Chong et al conducted a prospective cohort study of 31 patients who experienced at least 500mL blood loss during vaginal delivery. These investigators used POCUS to assess the IVC collapsibility index during the first, second, and third stages of labor as well as at the time of bleeding and following rapid resuscitation with 500mL of intravenous fluids. Chong and investigators then compared these indices to heart rate and mean arterial pressure at the same intervals and found that the IVC collapsibility index demonstrated more variation in response to volume status than did either heart rate or mean arterial pressure, both of which instead remained relatively stable over time. Moreover, a review of POCUS' role in monitoring the response to postpartum volume resuscitation was published in the American Journal of Obstetrics & Gynecology in 2024. This review suggested that the presence of three or more B-lines per screen on lung ultrasound is indicative of pulmonary edema during pregnancy and the postpartum period, as B-lines develop when air content in the lungs is replaced by transudate or exudate in the interstitium. It further suggested that an enlarged IVC diameter (> 2.0 cm) or minimal IVC collapsibility index (<15%) identified on POCUS could also be used to determine volume overload antenatally and postnatally.

The purpose of this study is to determine whether point-of-care ultrasound (POCUS) assessment of the lungs and inferior vena cava (IVC), both of which are a proxy for volume status, can be used to guide postpartum diuretic therapy in individuals with preeclampsia, and whether this strategy improves short-term maternal outcomes for this high-risk patient population.

The central study hypothesis is that, when guided by POCUS, use of diuretic therapy will improve postpartum outcomes in patients with preeclampsia relative to standard postpartum management alone. The investigators will test this hypothesis by conducting a pilot prospective cohort study that addresses the following aims:

Specific Aim 1: Assess the feasibility of POCUS assessment of the lungs and IVC in postpartum patients with preeclampsia within 24 hours of delivery.

To date, only a small handful of studies has evaluated the role of POCUS in patients with preeclampsia, the most recent of which was presented at the Society for Maternal-Fetal Medicine's Annual Pregnancy Meeting in February of this year. This pilot study conducted at the University of Tennessee Health Science Center compared the median IVC collapsibility index in 12 participants with preeclampsia with severe features to that in 10 participants without hypertensive disorders of pregnancy. Although the researchers found no significant difference in median IVC collapsibility index between the study groups, the results suggest that POCUS assessment of the IVC is at least feasible in a newly postpartum patient.

Thus, with respect to this specific aim, the investigators hypothesize that POCUS assessment will be able to successfully determine volume status in postpartum patients with preeclampsia. Specifically, the investigators anticipate that POCUS can be reliably used to identify the presence of B-lines in the lungs and to measure the greatest IVC diameter and IVC collapsibility index.

Specific Aim 2: Determine whether use of POCUS assessment to guide diuretic administration improves postpartum outcomes, including persistent hypertension at hospital discharge, time to normotension, antihypertensive use at hospital discharge, and hospital readmission, among patients with preeclampsia.

With respect to this specific aim, the investigators hypothesize that if oral or intravenous furosemide is administered to postpartum patients with preeclampsia following POCUS assessment that identifies 3 or more B-lines, an IVC diameter above 2cm, and/or an IVC collapsibility index less than 15%, there will be a decrease in persistent hypertension at hospital discharge (< 140/90 mm Hg and < 130/80 mm Hg), time to normotension, antihypertensive use at hospital discharge, and hospital readmission.

ELIGIBILITY:
Inclusion Criteria:

Historical cohort (group 1):

* Age greater than or equal to 18 years at the time of delivery
* Diagnosis of preeclampsia (without severe features, with severe features, HELLP syndrome, eclampsia) during pregnancy
* Gestational age greater than or equal to 20 weeks' gestation at delivery
* Delivery at the study institution within the 18-month period prior to implementation of the study's POCUS intervention
* Available and complete postpartum clinical data on: Daily blood pressure, diuretic or antihypertensive use, length of postpartum hospital stay, readmission within 30 days of primary hospitalization

Prospective cohorts (groups 2 and 3):

* Age greater than or equal to 18 years at the time of enrollment
* Diagnosis of preeclampsia (without severe features, with severe features, HELLP syndrome, eclampsia) made up until 24 hours postpartum Postpartum and within 24 hours of delivery

Exclusion Criteria:

Historical cohort (group 1):

* Delivery at an outside facility or incomplete postpartum records available for analysis
* Pre-existing diagnosis of chronic hypertension; selected to mirror prospective cohort exclusion criteria (see below).
* Documentation of chronic kidney disease (CKD stage 3 or higher); selected because diuresis is more likely to be avoided in this patient population even in the presence of physical exam findings suggesting volume overload.
* Documentation of postpartum complications unrelated to preeclampsia that may significantly alter hemodynamics (e.g., sepsis, postpartum hemorrhage); selected because diuresis is more likely to be avoided in this patient population even in the presence of physical exam findings suggesting volume overload.

Prospective cohorts (groups 2 and 3):

* Pre-existing diagnosis of chronic hypertension; selected because previous studies on furosemide use in patients with postpartum preeclampsia have found a significant reduction in hypertension among patients with newly diagnosed hypertensive disorders of pregnancy, but not among those with pre-gestational hypertension, meaning that inclusion of this population might reduce the magnitude of study effects.
* Baseline renal dysfunction with serum creatinine > 1.1 mg/dL; selected as this laboratory finding has been pre-selected as a safety outcome.
* Baseline hypokalemia with serum potassium < 3.5 mEq/L despite previous repletion with intravenous or oral potassium chloride; selected as this laboratory finding has been pre-selected as a safety outcome.
* Known hypersensitivity to furosemide or sulfa drugs; selected because this would preclude exposure to the study medication of interest.
* Current use of diuretics for other indications (e.g. heart failure); selected because this may require a furosemide or other diuretic regimen different from that planned for the study intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-06-15 (Estimated); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with persistent hypertension at time of postpartum hospital discharge | From study enrollment through completion of study participation, an average of 7 days or less
  Persistent hypertension at time of postpartum hospital discharge, defined both as blood pressure > 140/90 mm Hg according to American College of OB/GYN (ACOG) guidelines and 130/80 mm Hg according to Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (JNC-9) guidelines
Average days to resolution of hypertension | From study enrollment through completion of study participation, an average of 7 days or less
  Days to resolution of hypertension, defined both as blood pressure < 140/90 mm Hg according to ACOG guidelines and 130/80 mm Hg according to JNC-9 guidelines

SECONDARY OUTCOMES:
Proportion of subjects requiring antihypertensive medications at hospital discharge | From study enrollment through completion of study participation, an average of 7 days or less
  Need for antihypertensive medication at postpartum hospital discharge
Proportion of subjects requiring a secondary antihypertensive therapy at hospital discharge | From study enrollment through completion of study participation, an average of 7 days or less
  Addition of second antihypertensive agent during postpartum hospitalization
Average length of hospital stay | From birth through completion of study participation, an average of 7 days or less
  Length of postpartum hospitalization
Proportion of patients with a change in POCUS results over time | From study enrollment through completion of study participation, an average of 7 days or less
  Change in POCUS results from positive to negative for evidence of volume overload from the time of study enrollment through hospital discharge
Mean change in BNP levels over time | From study enrollment through completion of study participation, an average of 7 days or less
  Change in brain natriuretic peptide (BNP) levels from the time of study enrollment through hospital discharge
Proportion of patients with hospital readmission for high blood pressure | From time of initial hospital discharge through 30 days postpartum
  Readmission for blood pressure control within 30 days of discharge from initial postpartum hospitalization
Feasibility for future study | From study enrollment through completion of study participation, an average of 7 days or less
  Feasibility for future study, defined both as the number of subjects enrolled divided by the number of subjects with acceptable POCUS lung or IVC ultrasound images collected within 24 hours of delivery and as reliability between image assessment as performed by study staff and by blind reviewer

OTHER OUTCOMES:
Proportion of patients with hypotension | From study enrollment through completion of study participation, an average of 7 days or less
  Hypotension, defined as blood pressure < 90 mm Hg systolic and/or < 60 mm Hg diastolic
Proportion of patients with tachycardia | From study enrollment through completion of study participation, an average of 7 days or less
  Tachycardia, defined as heart rate > 100 beats per minute
Proportion of patients with moderate or severe hypokalemia | From study enrollment through completion of study participation, an average of 7 days or less
  Moderate or severe hypokalemia, defined as potassium < 3.0 mEq/L
Proportion of patients with acute kidney injury | From study enrollment through completion of study participation, an average of 7 days or less
  Acute kidney injury, defined as creatinine > 1.1 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Ashten B Waks, MD, MSPH, Principal Investigator — University of California, Irvine
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambrozic J, Brzan Simenc G, Prokselj K, Tul N, Cvijic M, Lucovnik M. Lung and cardiac ultrasound for hemodynamic monitoring of patients with severe pre-eclampsia. Ultrasound Obstet Gynecol. 2017 Jan;49(1):104-109. doi: 10.1002/uog.17331. Epub 2016 Dec 1. PMID 27736042
- [Background] Parra E, Brackney K, Piersall L, et al. (2025, January 26 - February 1). (1024) Comparing inferior vena cava collapsibility in postpartum patients with and without severe preeclampsia. Society for Maternal-Fetal Medicine 2025 Pregnancy Meeting, Denver, CO, United States.
- [Background] Gevaerd Martins J, Saad A, Saade G, Pacheco LD. The role of point-of-care ultrasound to monitor response of fluid replacement therapy in pregnancy. Am J Obstet Gynecol. 2024 Dec;231(6):563-573. doi: 10.1016/j.ajog.2024.06.039. Epub 2024 Jul 3. PMID 38969197
- [Background] Chong Y, Yu Y, Zhao Y, Zhang Y. Value of inferior vena cava diameter and inferior vena cava collapse index in the evaluation of peripartum volume: A prospective cohort study. Eur J Obstet Gynecol Reprod Biol. 2023 Jun;285:69-73. doi: 10.1016/j.ejogrb.2023.03.045. Epub 2023 Apr 11. PMID 37062116
- [Background] Lopes Perdigao J, Lewey J, Hirshberg A, Koelper N, Srinivas SK, Elovitz MA, Levine LD. Furosemide for Accelerated Recovery of Blood Pressure Postpartum in women with a hypertensive disorder of pregnancy: A Randomized Controlled Trial. Hypertension. 2021 May 5;77(5):1517-1524. doi: 10.1161/HYPERTENSIONAHA.120.16133. Epub 2021 Feb 8. PMID 33550824
- [Background] Ascarelli MH, Johnson V, McCreary H, Cushman J, May WL, Martin JN Jr. Postpartum preeclampsia management with furosemide: a randomized clinical trial. Obstet Gynecol. 2005 Jan;105(1):29-33. doi: 10.1097/01.AOG.0000148270.53433.66. PMID 15625138
- [Background] Balhotra K, Roach C, Al-Kouatly HB, Minkoff H, McLaren RA Jr. Association of antihypertensive medication at discharge with readmission for postpartum preeclampsia. Am J Obstet Gynecol. 2023 Jun;228(6):747-748.e1. doi: 10.1016/j.ajog.2023.01.020. Epub 2023 Jan 27. No abstract available. PMID 36716985
- [Background] Stevens W, Shih T, Incerti D, Ton TGN, Lee HC, Peneva D, Macones GA, Sibai BM, Jena AB. Short-term costs of preeclampsia to the United States health care system. Am J Obstet Gynecol. 2017 Sep;217(3):237-248.e16. doi: 10.1016/j.ajog.2017.04.032. Epub 2017 Jul 11. PMID 28708975
- [Background] Ditisheim A, Wuerzner G, Ponte B, Vial Y, Irion O, Burnier M, Boulvain M, Pechere-Bertschi A. Prevalence of Hypertensive Phenotypes After Preeclampsia: A Prospective Cohort Study. Hypertension. 2018 Jan;71(1):103-109. doi: 10.1161/HYPERTENSIONAHA.117.09799. Epub 2017 Nov 13. PMID 29133363
- [Background] Gestational Hypertension and Preeclampsia: ACOG Practice Bulletin, Number 222. Obstet Gynecol. 2020 Jun;135(6):e237-e260. doi: 10.1097/AOG.0000000000003891. PMID 32443079

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT07167862/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT07167862/ICF_001.pdf